CLINICAL TRIAL: NCT01182337
Title: A Multicenter, Randomized, Double-blind, Placebo Controlled, Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Effectiveness of Single Administration Intradiscal rhGDF-5 for the Treatment of Early Stage Lumbar Disc Degeneration
Brief Title: A Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Effectiveness of Single Administration Intradiscal rhGDF-5 for the Treatment of Early Stage Lumbar Disc Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DePuy Spine (Industry)
Collaborators: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 09-Intradiscal rhGDF-5-03
Record Dates: First submitted 2010-08-11; First posted 2010-08-16 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Early Lumbar Disc Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intradiscal rhGDF-5 (Experimental): The API is recombinant human growth and differentiation factor-5 (rhGDF-5), a recombinant version of human GDF-5. GDF-5 is a member of the transforming growth factor-b (TGF-b) superfamily and the bone morphogenetic protein (BMP) subfamily, and is known to influence the growth and differentiation of various tissues, including the intervertebral disc. In vitro experiments have shown that rhGDF-5 can stimulate gene expression and synthesis of the extracellular matrix proteins type II collagen and aggrecan. In vivo experiments in rabbit models of disc degeneration have shown that intradiscal injections of rhGDF-5 can stimulate an increase in disc height and hydration.
  Interventions: Drug: Intradiscal rhGDF-5
- Vehicle control (Placebo Comparator): Excipients in Intradiscal rhGDF-5, to include Trehalose, Glycine, HCl, and Water for Injection
  Interventions: Drug: Vehicle control

INTERVENTIONS:
Drug: Intradiscal rhGDF-5 — The API is recombinant human growth and differentiation factor-5 (rhGDF-5), a recombinant version of human GDF-5. GDF-5 is a member of the transforming growth factor-b (TGF-b) superfamily and the bone morphogenetic protein (BMP) subfamily, and is known to influence the growth and differentiation of various tissues, including the intervertebral disc. In vitro experiments have shown that rhGDF-5 can stimulate gene expression and synthesis of the extracellular matrix proteins type II collagen and aggrecan. In vivo experiments in rabbit models of disc degeneration have shown that intradiscal injections of rhGDF-5 can stimulate an increase in disc height and hydration.
  Arms: Intradiscal rhGDF-5
Drug: Vehicle control — Excipients in Intradiscal rhGDF-5, to include Trehalose, Glycine, HCl, and Water for Injection
  Arms: Vehicle control

SUMMARY:
Study to show the safety, tolerability and preliminary effectiveness of Intradiscal rhGDF-5 in subjects with early lumbar disc degeneration

ELIGIBILITY:
Inclusion Criteria:

1. Persistent low back pain with at least 3 months of non-surgical therapy at one suspected symptomatic lumbar level (L3/L4 to L5/S1) as confirmed using a standardized discography protocol. The required discography protocol will be provided by the sponsor. Subjects with multilevel disease must have a provocative discogram confirming that only 1 level is symptomatic at least 2 weeks prior to administration, with an expiry of 12 months from the date performed.
2. Oswestry Disability Index (ODI) for low back pain of 30 or greater
3. Low Back Pain score greater than or equal to 4 cm as measured by Visual Analog Scale (VAS) at Visit 1 Baseline
4. Male or Female 18 years of age or older

Exclusion Criteria:

1. Persons unable to have a discogram, CT, or MRI
2. Abnormal neurological exam at baseline (e.g., chronic radiculopathy)
3. Active radicular pain due to anatomical compression such as stenosis or disc herniation (radicular pain is defined as pain below the knee)
4. Extravasation of contrast agent during the discogram into the epidural space (does not include leakage of contrast agent along the needle track or leakage to the outer annular ring at the posterior longitudinal ligament vicinity)
5. Suspected symptomatic facet joints and/or severe facet joint degeneration at the index level or adjacent segments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Yeungnam University Medical Center, Daegu
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary Hospital, Seoul
  - Yonsei University Health System, Seoul

REFERENCES:
- [Derived] Adoungotchodo A, Epure LM, Mwale F, Lerouge S. Chitosan-based hydrogels supplemented with gelatine and Link N enhance extracellular matrix deposition by encapsulated cells in a degenerative intervertebral disc environment. Eur Cell Mater. 2021 May 4;41:471-484. doi: 10.22203/eCM.v041a30. PMID 33945627

RESULTS

PARTICIPANT FLOW:
Groups:
- Intradiscal rhGDF-5 1.0mg: The API is recombinant human growth and differentiation factor-5 (rhGDF-5), a recombinant version of human GDF-5. GDF-5 is a member of the transforming growth factor-b (TGF-b) superfamily and the bone morphogenetic protein (BMP) subfamily, and is known to influence the growth and differentiation of various tissues, including the intervertebral disc.
Period: Overall Study
Arm/Group | Intradiscal rhGDF-5 1.0mg | Vehicle Control
Started | 22 | 9
Completed | 19 | 7
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intradiscal rhGDF-5: The API is recombinant human growth and differentiation factor-5 (rhGDF-5), a recombinant version of human GDF-5. GDF-5 is a member of the transforming growth factor-b (TGF-b) superfamily and the bone morphogenetic protein (BMP) subfamily, and is known to influence the growth and differentiation of various tissues, including the intervertebral disc.
- Total: Total of all reporting groups
Arm/Group | Intradiscal rhGDF-5 | Vehicle Control | Total
Number analyzed (Participants) | 22 | 9 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (11.78) | 40.6 (15.63) | 41.2 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 12 | 6 | 18
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 22 | 9 | 31

OUTCOME MEASURES:

1. Primary Outcome: Neurological Assessment for Motor Function and Reflexes/Sensory
Description: Neurological Assessment for Motor Function and Reflexes/Sensory- Number of patients with Clinically Significant Abnormal results at 12 months.
  For Motor Function, Clinically Significant Abnormal results are determined by the surgeon investigator and are further classified by grade: 0= No Movement, 1= Flicker/trace of contraction, 2=Active movement when gravity removed, 3= Active movement against gravity, 4= Active Movement against gravity and resistance.
  For Reflexes/Sensory, Clinically Significant Abnormal results are determined by the surgeon investigator and are based on exams of the Knee, Ankle, L3-L5 Dermatone, and S1 Dermatome. Tension signs are evaluated with a straight leg raise to determine at which point, if any, sciatic pain occurs.
Time Frame: 12 months
Population: Safety Population
  For the Neurological Assessment at 12 months, only 21 subjects from the rhGDF-5 group completed the assessment (out of 22 total subjects) and 5 subjects from the Control group completed the assessment (out of 9 subjects total).
Measure: Number; unit: participants
Arm/Group | Intradiscal rhGDF-5 1.0mg | Vehicle Control
Number analyzed (Participants) | 21 | 5
participants | 0 | 0

2. Secondary Outcome: Change in Function Assessed by Oswestry Disability Index Change at 12 Months From Baseline.
Description: The Oswestry Disability Index (ODI) is a 10-category (Pain Intensity, Personal Care, Lifting, Walking, Sitting, Standing, Sleeping, Sex Life, Social Life, Traveling) disability measurement scale with a graded response from 0 to 5, with 0 being the best score (no impairment) to 5 being the worst score (significant impairment). ODI score for a subject is calculated by adding the scores and converting the score to a 100 point scale.
Time Frame: 12 month
Population: FAS Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 1.0mg | Vehicle Control
Number analyzed (Participants) | 22 | 9
units on a scale | -13.5 (13.86) | -10.4 (8.98)

3. Primary Outcome: Treatment Emergent Adverse Events- Relationship to Study Drug
Description: Number of patients with Treatment Emergent Adverse Events that were designated as Definitely Related to Study Drug.
Time Frame: Through a 12 month period and annual telephone contact at 24 and 36 months for subject health status follow-up
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Intradiscal rhGDF-5 1.0mg | Vehicle Control
Number analyzed (Participants) | 22 | 9
participants | 0 | 0

4. Primary Outcome: Treatment Emergent Adverse Events- Relationship to Study Drug
Description: Number of patients with Treatment Emergent Adverse Events that were designated as Possibly or Probably Related to Study Drug.
Time Frame: 12 month period and annual telephone contact at 24 and 36 months for subject health status follow-up
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Intradiscal rhGDF-5 | Vehicle Control
Number analyzed (Participants) | 22 | 9
participants | 0 | 1

5. Secondary Outcome: Change in Pain Visual Analog Scale (VAS) at 12 Months From Baseline.
Description: The Visual Analog Scale (VAS) pain score asks the subject to place a vertical mark on a horizontal line (that is approximately 10 cm long) with 'No Pain' (score of 0 = 0 cm) listed on the left and 'Very severe pain' (score of 10=10cm) labeled on the right. The subject is instructed to indicate the amount of pain they feel in their back.
Time Frame: 12 months
Population: FAS Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 1.0mg | Vehicle Control
Number analyzed (Participants) | 22 | 9
units on a scale | -2.49 (2.211) | -1.42 (3.177)

6. Secondary Outcome: Change in Physical Component Summary of Quality of Life Measure Assessed by Short Form 36 at 12 Months From Baseline
Description: The 36-item Short Form Health Survey (SF-36) is a patient reported outcome survey that evaluates functional health and well-being. The survey is converted into two summary measures (the Physical Component - PCS and Mental Component- MCS) that are scored from 0 to 100 (where 100 indicates the highest level of health).
Time Frame: 12 months
Population: FAS Population
  Only 21 subjects from the rhGDF-5 group (out of 22 total subjects) completed the baseline PCS, SF-36.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 1.0mg | Vehicle Control
Number analyzed (Participants) | 21 | 9
units on a scale | 2.52 (7.354) | 3.24 (9.879)

7. Secondary Outcome: Change in Mental Component Summary Quality of Life Measure Assessed by Short Form SF-36 at 12 Months From Baseline.
Description: as for outcome 6
Time Frame: 12 Months
Population: FAS Population
  Only 21 subjects from the rhGDF-5 group (out of 22 subjects total) completed the MCS, SF-36.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 1.0mg | Vehicle Control
Number analyzed (Participants) | 21 | 9
units on a scale | 4.03 (14.050) | 4.34 (10.727)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through a 12 month period and annual telephone contact at 24 months and 36 months
Arm/Group | Intradiscal rhGDF-5 | Vehicle Control
Serious Adverse Events (participants affected / at risk) | 5/22 | 2/9
Other Adverse Events (participants affected / at risk) | 16/22 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intradiscal rhGDF-5 (N=22) | Vehicle Control (N=9)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intradiscal rhGDF-5 (N=22) | Vehicle Control (N=9)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 3 (4)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Varicose Vein (Vascular disorders) | 0 (0) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (3) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Investigators may freely present or publish results of the Clinical Investigation in a manner which fairly sets forth the conclusions reached by the Clinical Investigators, but only after the Sponsor has been given the opportunity of reviewing the proposed presentation or publication at least 60 days prior to the intended submission, presentation, or publication date.